CLINICAL TRIAL: NCT00477243
Title: Locus of Control and Spirituality in Palliative Care Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2003-1044; NCI-2010-00593 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Palliative Care Patients; Spirituality; Locus of Control; Questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palliative Care Clinic Patients: Department of Symptom Control and Palliative Care Center Patients
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 8 questionnaires will take about 40 minutes to complete.

SUMMARY:
Primary Objectives:

1. To determine whether the degree of spirituality/religiosity as determined by the Duke University Religion Index and Functional Assessment of Chronic Illness Therapy-Spiritual Well Being Scale (FACIT-Sp) correlates with internal locus of control as determined by the Locus of Control Scale.
2. To determine the relationships among spiritual-well being, religiosity, hope, depression, and culture, socioeconomic status, and gender in a palliative care setting.
3. To determine if hope and depression in palliative care patients are affected by the degree of intrinsic and extrinsic spirituality/religiosity.
4. To determine if patients who believe in predestination correlate with decreased locus of control, but improved quality of life and degree of religiosity.

DETAILED DESCRIPTION:
If you are receiving care in the Palliative Care clinic and are eligible to participate, you will be asked to fill out one-time quality of life surveys, which will take about 40 minutes to complete. The Functional Assessment of Chronic Illness Therapy (FACT-G) survey asks questions about physical and emotional well-being, functional well-being (how much you participate in and enjoy normal daily activities), and social/family well-being.

This study first collected questionnaires from 100 participants from different racial and ethnic backgrounds. When the questionnaires were compared, investigators found some interesting differences between the African American and Caucasian participants. To better understand these findings, an additional 67 African American patients are needed to compare the groups.

The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACT-Sp) asks questions about personal meaning, faith and peace. The Duke University Religion Index (DUREL) asks questions about religious practices. The Locus of Control (LOC) questionnaire asks questions about personal internal control, your views on chance, and your views on power. The Herth Health Scale (HHS) asks questions about hope. The Edmonton Symptom Assessment System (ESAS) asks questions about symptoms you may be experiencing. The Hospital Anxiety and Depression Scale (HADS) asks questions about your feelings of depression and anxiety. The "predetermination" questionnaire asks questions about your beliefs about your fate.

These eight questionnaires will take about 40 minutes to complete and may be completed at a later time if you become tired. Information about you will also be collected (such as your age and gender).

This is an investigational study. About 167 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 17 years (surveys have not been validated in minors)
2. Expected survival > 6 weeks
3. Patients experiencing acute side effects from chemotherapy (mucositis, emesis, or severe grade 2-3 neuropathy) are not eligible
4. No clinical evidence of cognitive failure, with normal Mini Mental State Examination (MMSE). A score of 24 is considered normal
5. Only new patients presenting to the Department of Symptom Control and Palliative Care Center

Exclusion Criteria:

1) N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Symptom Control and Palliative Care at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-06-03 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-11 (Actual)

PRIMARY OUTCOMES:
Determination of Spirituality/Religiosity in Correlation With Internal Locus of Control. | 40 minutes to complete questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org